CLINICAL TRIAL: NCT00316576
Title: Evaluation of the Impact of the Angiotensin-Converting Enzyme Insertion/Deletion Polymorphism on the Development of Acute Renal Failure in Critically Ill Patients
Brief Title: Angiotensin-Converting Enzyme Polymorphism and Acute Renal Failure (ECAREA)
Status: Terminated | Type: Observational
Why Stopped: The study was stopped on november 2006 after inclusion was fulfilled
Sponsor: University Hospital, Caen (Other)
Other Study IDs: 05-130
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Kidney Failure, Acute; Critical Illness
Keywords: Kidney failure, Acute; Genetic Polymorphism; Angiotensin-converting enzyme
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness | interventions — Blood Specimen Collection; Polymerase Chain Reaction

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Blood sampling for PCR

SUMMARY:
Associations between angiotensin-converting enzyme gene polymorphism and occurrence and outcome of ARDS, and with respiratory complications post cardiopulmonary bypass have already been demonstrated. Based on physiological effects of angiotensin II, we hypothesized that the I allele of the angiotensin-converting enzyme Insertion/Deletion polymorphism may be associated with a higher risk of acute renal failure in critically ill patients.

DETAILED DESCRIPTION:
Associations between angiotensin-converting enzyme gene polymorphism and occurrence and outcome of ARDS, and with respiratory complications post cardiopulmonary bypass have already been demonstrated. Based on physiological effects of angiotensin II, we hypothesized that the I allele of the angiotensin-converting enzyme Insertion/Deletion polymorphism may be associated with a higher risk of acute renal failure in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs
* ICU stay > 48 hours

Exclusion Criteria:

* Age < 18 yrs
* Creatinine > 180 µmol/L
* Absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to ICU fore more than 48 hours
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2006-05; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Incidence of ARF | During ICU stay

SECONDARY OUTCOMES:
Mortality | ICU and Hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Damien du Cheyron, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Medical Intensive care Unit; Caen University Hospital, Caen, France

REFERENCES:
- [Derived] du Cheyron D, Fradin S, Ramakers M, Terzi N, Guillotin D, Bouchet B, Daubin C, Charbonneau P. Angiotensin converting enzyme insertion/deletion genetic polymorphism: its impact on renal function in critically ill patients. Crit Care Med. 2008 Dec;36(12):3178-83. doi: 10.1097/CCM.0b013e318186a299. PMID 19020433